CLINICAL TRIAL: NCT03397251
Title: Dissected Aorta Repair Through Stent Implantation (DARTS): A Feasibility, Safety and Performance Trial
Brief Title: DARTS I: Feasibility, Safety, and Performance Trial
Acronym: DARTS I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascyrus Medical LLC. (Industry)
Collaborators: Artivion Inc. (Industry)
Responsible Party: Sponsor
Organization: Artivion Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DARTS-AMDS
Record Dates: First submitted 2018-01-06; First posted 2018-01-11 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Acute DeBakey I Aortic Dissection; Intramural Hematoma

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, non-blinded, single-arm study evaluating the feasibility and safety of the AMDS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AMDS Implantation (Experimental): AMDS implantation is performed during an open chest procedure for intervention of aortic dissection repair.
  Interventions: Device: AMDS

INTERVENTIONS:
Device: AMDS — The device will be implanted during an already planned surgical intervention for aortic dissection repair. The participant will be observed and data gathered during the surgery and routine standard of care follow up visits.

SUMMARY:
The objective of this study is to investigate the feasibility and clinical benefits of the AMDS to treat patients with acute DeBakey type I dissections and/or intramural hematomas (IMH) involving the ascending aorta and aortic arch through open surgical repair.

DETAILED DESCRIPTION:
AMDS is designed to complement the replacement of the ascending aorta with conventional surgical technique utilizing a conventional polyester graft. AMDS is constructed of an uncovered Nitinol wire braided stent attached proximally to a polytetrafluoroethylene (PTFE) felt graft component. The PFTE felt graft component excludes the FL at the distal aortic anastomosis and the wire stent re-expands the dissection flap within the arch and descending aorta, which aims to treat malperfusion and promote positive remodeling of the aorta.

The DARTS I Feasibility, Safety and Performance trial is a prospective, non-randomized, non-blinded, single-arm, multi-institutional Canadian study evaluating the feasibility and safety of the AMDS graft. A goal of 30 subjects will be enrolled at 1 site in Germany.

The enrollment period will span a minimum of 3 months from Institutional Review Board (IRB) approval and site activation. Candidates for this study are adults who require repair of an acute DeBakey type I aorta dissection and/or intramural hematoma (IMH). Patients will be consented pre-operatively and enrolled patients will be followed for approximately 5 years after their AMDS implantation date. Data will be collected at 10 time points: baseline (pre-operatively), discharge, 1 month post-operatively, 3 months post-operatively, and 6 months post-operatively, 1 year post-operatively and thereafter, annually, for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent obtained
2. ≥18 years of age or ≤80 years of age (male or female)

   Subject must have one of the following diagnosed, based on CT angiography, within 0-14 days:
3. Acute DeBakey I dissection or
4. Acute DeBakey I intramural hematoma (IMH)

Exclusion Criteria:

General Exclusion Criteria

Patients must be excluded from the study if any of the following conditions are true:

1. Less than 18 years of age or over 80 years of age
2. Life expectancy less than 2 years
3. Pregnant or breastfeeding or planning on becoming pregnant within 60 months
4. Unwilling to comply with the follow-up schedule
5. Refusal to give informed consent
6. Institutionalized individualized due to administrative or judicial order
7. Individuals with a dependent relationship to the sponsor or investigator

Medical Exclusion Criteria

Patients must be excluded from the study if any of the following conditions are true:

1. Uncontrolled systemic infection
2. Uncontrollable anaphylaxis to iodinated contrast
3. Known allergy(ies) to Nitinol and/or PTFE
4. Patient in extreme hemodynamic compromise requiring cardiopulmonary resuscitation (CPR)
5. Inability to obtain CT angiograms for follow-up
6. Previously diagnosed with Marfan syndrome, Loeys- Dietz syndrome or Ehlers- Danlos syndrome with confirmed laboratory genetic testing on a date prior to the diagnosis of the dissection

Anatomical Exclusion Criteria

1. Any pathology of mycotic origin
2. Subacute or chronic dissection of the ascending aorta and aortic arch (>14 days after the index event)
3. Aortic fistulous communication with non-vascular structure (e.g. esophagus, bronchial)
4. Extensive thrombus or calcifications in the aortic arch as defined by CT angiography
5. Excessive tortuosity precluding safe passage of the AMDS as defined by CT angiography
6. Descending thoracic aneurysm involving the proximal third (1/3) of the descending aorta and measuring > 45mm in diameter
7. Aortic arch aneurysm > 45mm in diameter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related mortality | 12 weeks
  The number of patients with mortality related to the treatment device
Number of participants with treatment-related neurological deficit | 12 weeks
  The number of patients with neurological complications related to the treatment device
Number of patients with aortic injury associated with the implantation of the device | 12 weeks
  The number of patients with aortic injury related to the treatment device
Aortic arch branch vessel patency | 12 weeks
  The number of patients with arch branch vessel stenosis/ occlusion related to the treatment device

SECONDARY OUTCOMES:
Number of participants with treatment-related mortality | 24 weeks and 12 months
  The number of patients with mortality related to the device and procedure
Number of participants with treatment-related neurological deficit | 24 weeks and 12 months
  The number of patients with neurological complications, such as stroke, TIA, and paralysis/paraplegia) related to the treatment device
Number of patients with aortic injury associated with the implantation of the device | 24 weeks and 12 months
  The number of patients with aortic injury related to the treatment device
Aortic arch branch vessel patency | 24 weeks and 12 months
  The number of patients with arch branch vessel stenosis/ occlusion related to the treatment device

OTHER OUTCOMES:
Re-expansion of the true lumen | 12 weeks, 24 weeks, and 12 months
  The number of patients with achieved re-expansion of the true lumen following AMDS implantation
False lumen reattachment/positive remodeling | 12 weeks, 24 weeks, and 12 months
  The number of patients which exhibit positive remodeling/false lumen reattachment as measured by CT.
False Lumen Thrombosis | 12 weeks, 24 weeks, and 12 months
  The percentage of patients with evidence of false lumen thrombosis within the confinement of the AMDS, distal to the AMDS but proximal to the Celiac trunk, along the paravisceral aorta and in the infrarenal aorta.
Stent-graft integrity Assessment | 12 weeks, 24 weeks, and 12 months
  The percentage of patients without evidence of stent-graft fractures, kinking, or twisting leading to occlusion or ischemia in patients that have undergone aortic dissection repair with AMDS. Stent graft integrity will be evaluated by CTA with a Core Imaging Lab.
Successful device deployment | 12 weeks, 24 weeks, and 12 months
  The number of patients which had successful device deployment
AMDS removal | 12 weeks, 24 weeks, and 12 months
  The percentage of patients that required AMDS removal
AMDS related re-interventions after the dissection repair | 12 weeks, 24 weeks, and 12 months
  The percentage of patients with need of secondary intervention related to the AMDS implantation following the index procedure for aortic dissection repair
Cardiopulmonary bypass (CBP) duration | 12 weeks, 24 weeks, and 12 months
  The total time (in minutes) of CBP required for patients undergoing AMDS implantation
Circulatory arrest duration | 12 weeks, 24 weeks, and 12 months
  The total time (in minutes) of circulatory arrest for patients undergoing AMDS implantation
Time in ICU | 12 weeks, 24 weeks, and 12 months
  The total amount of days for patients that have undergo aortic dissection repair with AMDS implantation
Duration of hospitalization | 12 weeks, 24 weeks, and 12 months
  The total number of days of hospitalization required for patients undergoing AMDS implantation
AMDS procedure duration | 12 weeks, 24 weeks, and 12 months
  The total amount of time (in minutes) that it takes for AMDS to be implanted

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Kempfert, MD, Principal Investigator — German Heart Institute
Locations (1):
- Deutsches Hertzzentrum Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montagner M, Kofler M, Heck R, Buz S, Starck C, Kurz S, Falk V, Kempfert J. Initial experience with the new type A arch dissection stent: restoration of supra-aortic vessel perfusion. Interact Cardiovasc Thorac Surg. 2021 Jul 26;33(2):276-283. doi: 10.1093/icvts/ivab085. PMID 34010408
- [Background] Bozso SJ, Nagendran J, Chu MWA, Kiaii B, El-Hamamsy I, Ouzounian M, Kempfert J, Starck C, Moon MC. Midterm Outcomes of the Dissected Aorta Repair Through Stent Implantation Trial. Ann Thorac Surg. 2021 Feb;111(2):463-470. doi: 10.1016/j.athoracsur.2020.05.090. Epub 2020 Jul 13. PMID 32673661
- [Background] Bozso SJ, Nagendran J, Chu MWA, Kiaii B, El-Hamamsy I, Ouzounian M, Kempfert J, Starck C, Shahriari A, Moon MC. Single-Stage Management of Dynamic Malperfusion Using a Novel Arch Remodeling Hybrid Graft. Ann Thorac Surg. 2019 Dec;108(6):1768-1775. doi: 10.1016/j.athoracsur.2019.04.121. Epub 2019 Jun 27. PMID 31254509